CLINICAL TRIAL: NCT05860829
Title: Effect of Nutrition and Oral Hygiene Education Using Telehealth on Diet Diversity, Nutrition Literacy and Oral Hygiene Practices in Children With Autism: A Mixed-method Stud
Brief Title: Effect of Nutrition and Oral Hygiene Education Using Telehealth on Diet Diversity, Nutrition Literacy and Oral Hygiene Practices in Children With Autism: A Mixed-method Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Aliya Haider, Principal Investigator, Dow University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DowUniHS
Record Dates: First submitted 2023-05-06; First posted 2023-05-16 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Oral hygiene; Nutrition literacy; Diet Diversity; Caregiver's experience; Telehealth; Caregiver
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: A pre-test will be conducted to explore the level of knowledge of the caregivers regarding oral hygiene and nutrition literacy of children with ASD. In-depth interviews will be conducted in order to identify the problems faced by caretakers till the saturation is reached. A semi-structured interview guide and caregiver education program will be developed related to dietary intake and oral hygiene of the child with autism for the caregivers. A dentist will provide education on oral hygiene and a registered dietician on nutrition literacy and diet diversity via telehealth. A post-test will be conducted after completion of all the sessions to assess the impact of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Caregivers of children with Autism Spectrum Disorder (ASD) (Experimental): Arm includes only the caregivers of children with ASD. The knowledge of caregivers of children with ASD regarding oral and nutritional health and the burdens they encounter in dealing and caring for these children will be assessed. Then, educating caregivers on diet diversities, and effective oral health education, expecting from it to the eating habits and oral hygiene of children living with autism.
  Interventions: Behavioral: Educational

INTERVENTIONS:
Behavioral: Educational — Caregivers of children with ASD will be sampled that are enrolled in Autism specialized Schools or centers. Tools and group education sessions will be developed in Urdu, English and Sindhi language. A caregiver education program session will be conducted by a practicing dentist and a registered dietitian in Urdu1 and English. Considering the ease of caregivers, cost-effectiveness and managing flexible hours, tele-health will be practiced for education program. A post-test will be conducted to assess the impact of the educational program on the knowledge of caregivers.

SUMMARY:
The goal of this interventional study is to assess the knowledge of caregivers of children with Autism Spectrum Disorder (ASD) regarding oral and nutritional health and the burdens they encounter in dealing and caring for these children. The main aims to answer are:

Educating caregivers on

* Diet diversities
* Improving oral health habits Participants will have to
* Fill questionnaires
* Undergo educational sessions
* Fill post education questionnaires Researchers will compare pre and post educational questionnaires to see if the intervention makes a difference.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder defined by deficits in social communication and the presence of restricted and repetitive behaviors and interests. The disorder incorporates the constraints and typical behaviors in early childhood, which later becomes problematic to function in society. Although the reason of ASD are unexplained yet, however, air pollution, organic toxicants, seasonal factors, psychological stress, migration, birth order and nutrition may have a close relationship with the incidence of ASD. Emphasizing on the fact that it is a lifelong condition and there is no specific cure to it, it can only be managed and assisted by caregivers specially. Every individual with ASD have a unique and different behavioral pattern. These behavioral patterns are managed by experts of behavior management such as speech or occupational therapists.

Poor oral hygiene is widely reported among children with autism, thus can elevate the likelihood of dental cavities and bad breath. Dental health can be further deteriorated if a child with ASD prefers soft, sweet and sticky food preferences as unhealthy diet intake and limited diet diversity. Food selectivity and other feeding problems are endemic in children with autism spectrum disorders (ASD).

In Pakistan, few studies have comprehensively looked at the children with special needs.

As Pakistan is a Low-Middle-Income country (LMIC) with limited sources and ASD is a domain that still needs more research work to be done. There is a majority of population that overlook the topic and then there is a category that strongly believes myths and misconceptions that evolve regarding 'treatment' and management of Autism in individuals. Another setback is a limited number Professionals with sound knowledge of the disorder that can cater to majority individuals and their caregivers, providing assistance in how to manage the most basic things like oral hygiene and nutritional education - that can ultimately encourage the reduction of burden in caregivers.

ELIGIBILITY:
Inclusion Criteria:

1. Caregivers of Children (5-18 years) with Autism enrolled in Autistic or specialized Schools.
2. Caregivers able to communicate in English or Urdu or Sindhi.
3. Caregiver of one child with Autism.
4. Caregivers with smartphone/laptop/IPhone and internet facility.

Exclusion Criteria:

1. Caregiver of child with Autism living with any known food allergies.
2. Caregiver of child with Autism enrolled in any other trial.
3. Caregiver of child with Autism and any other mental disorders.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 123 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-08-03 (Actual); Study Completion 2024-09-21 (Actual)

PRIMARY OUTCOMES:
Effect of nutrition education on nutrition literacy | Including pre test, intervention and post test - will require 6 months (roughly).
  Nutrition literacy Assessment Instrument (NLit) will be used to assess the nutrition literacy.
Effect of nutrition education on diet diversity | Including pre test, intervention and post test - will require 6 months (roughly).
  Diet Diversity Score (DDS) will be used to assess diet diversity. There are twelve questions in this questionnaire. The number of food groups consumed by the child from the total number of twelve food groups will either be '0' or '1' which will be summed up. The scoring will be done, low will be ≤ 4 food groups, medium will be considered as 5 to 8 food groups, and high will be 9 to 12 food groups.
Effect of oral hygiene education on oral hygiene practices. | Including pre test, intervention and post test - will require 6 months (roughly).
  Oral hygiene assessment score will be used to assess oral hygiene practices. There are a total of ten questions in this section. The interpretation will be done with the help of pre oral hygiene education and post oral hygiene education and the difference it creates among the caregivers of children with Autism.

SECONDARY OUTCOMES:
Assessment of experience of caregivers of children with Autism | Including pre test, intervention and post test - will require 6 months (roughly).
  Caregiver burden assessment scoring will be done by COPE Index. COPE index is a 15 item questionnaire developed to assess the caregiver experiences. Questions cover negative, positive and social aspects of caregiving. Score above 12 is for Negative Impact or below 12 for Positive Value.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Effort Welfare Trust, Karachi, Sindh
  - Markaz e Umeed, Karachi, Sindh